CLINICAL TRIAL: NCT00254618
Title: Study to Determine the Pharmacokinetics of Mesalamine Following Administration of 30, 60, and 90 mg/kg/Day as 400 mg Delayed-release Tablets Given Every 12 Hours for 28 Days to Children/Adolescents With Active Ulcerative Colitis.
Brief Title: A Study of Asacol Absorption, Metabolism and Excretion in Children and Adolescents With Ulcerative Colitis.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment.
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2005018
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; pharmacokinetics; pediatrics
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 30 mg (Experimental): 30 mg/kg/day mesalamine
  Interventions: Drug: mesalamine
- 60 mg (Experimental): 60 mg/kg/day mesalamine
  Interventions: Drug: mesalamine
- 90 mg (Experimental): 90 mg/kg/day mesalamine
  Interventions: Drug: mesalamine

INTERVENTIONS:
Drug: mesalamine — oral tablet, 30 mg mesalamine/day for 28 days
  Arms: 30 mg
Drug: mesalamine — oral tablet, 60 mg mesalamine/day for 28 days
  Arms: 60 mg
Drug: mesalamine — oral tablet, 90 mg mesalamine/day for 28 days
  Arms: 90 mg

SUMMARY:
The purpose of this randomized, open-label, parallel-group study is to determine how the body absorbs and eliminates mesalamine following administration of either 30 mg/kg/day, 60 mg/kg/day or 90 mg/kg/day as 400 mg delayed-release tablets given every 12 hours of 28 days to children and adolescents with active ulcerative colitis.

DETAILED DESCRIPTION:
Ulcerative colitis is a type of inflammatory bowel disease characterized by diffuse, continuous inflammation of the colon. Recent estimates suggest that approximately 17,000 children between 5 and 17 years of age in the U.S. are diagnosed with ulcerative colitis. Estimates of average age at onset in children vary, although 80-90% of patients are 9 years of age or older when symptoms develop.

Asacol is a delayed-release tablet formulation designed to deliver mesalamine (also known as mesalazine) at a pH ≥ 7.0. This property results in release of the drug in the terminal ileum and beyond. Physiologic factors such as the pH of the surrounding medium, transit times in the intestinal regions of interest, and the rate and extent of absorption and metabolism govern Asacol drug release and delivery, which in turn influence the pharmacokinetic profile of the delivered drug. These physiologic factors and their effect on Asacol pharmacokinetics have been studied in adults, but corresponding studies in children have not been performed. However, relevant studies describing the gastrointestinal pH; transit times; and pharmacokinetic aspects of drug absorption, metabolism, and excretion in pediatric patients (relative to adults) provide reasons to expect that the performance characteristics of Asacol in the pediatric population will be similar to those measured in adults.

In a compassionate-use study that included 66 children between the ages of 3 and 16 years, the safety profile of long-term mesalamine therapy (10 to 93 mg/kg/day) was similar to that observed among adult patients enrolled in the study. In addition, in a retrospective study of 732 pediatric patients with inflammatory bowel disease (153 of whom were treated with mesalamine), D'Agata, et al. concluded that mesalamine was safe and well tolerated when used long term at doses ranging from 13 to 111 mg/kg/day. Although few clinical studies of mesalamine have been performed in children, pediatric gastroenterologists use mesalamine to treat children with inflammatory bowel disease, and doses higher than those proposed for this study (up to 100 mg/kg/day) have been recommended.

This study will provide information about the pharmacokinetics of mesalamine and its major metabolite in children being treated with Asacol for mildly to moderately active ulcerative colitis. It was designed to meet the expectations outlined in a Written Request issued by the FDA, as well as regulatory requirements to study the weight-based equivalent of 4.8 g/day. The age-appropriate dose formulation, the 400 mg tablet, will be used, and patients will be dosed every 12 hours, since this regimen is considered more convenient for pediatric patients and their parents.

During this open-label, randomized, 4-week parallel-group study in pediatric patients, patients will be stratified by age (5-8 years and 9-17 years), and randomly assigned to one of 3 dose levels (30 mg/kg/day, 60 mg/kg/day, and 90 mg/kg/day) in the manner described in Section 3.5.1. Patients weighing less than 20 kg will not be assigned to the 30 mg/kg group, and patients weighing more than 60 kg will not be assigned to the 90 mg/kg group, due to dosing concerns. A total of 48 patients will be enrolled (8/treatment group/age stratum), with the expectation that 36 (6/treatment group/age stratum) will complete.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to participate in the study if they have/are:

1. male or female between the ages of 5 and 17 years, inclusive, at the time of the first dose of study medication
2. mildly to moderately active ulcerative colitis (either newly- or previously-diagnosed), as confirmed by their physician, for which mesalamine would be used as part of their normal treatment
3. generally in good health (other than the diagnosis of ulcerative colitis), based on medical history, physical examination, and screening laboratory results
4. able to swallow Asacol tablets (400 mg marketed US formulation)
5. a body weight no less than 16 kg and no more than 90 kg
6. able and willing to participate in the study and follow study procedures, as evidenced by providing assent and having a parent/guardian-signed written informed consent.

Exclusion Criteria:

Patients will be excluded from the study if they have/are:

1. a history of cancer 2. a history of intestinal surgery or malabsorption 3. a history of renal insufficiency 4 a history of allergy or hypersensitivity to salicylates or aminosalicylates 5. evidence of clinically significant organic or psychiatric disease on medical history or physical examination that, in the Investigator's opinion, would prevent the patient from completing the study or would jeopardize the patient's safety 6. a creatinine clearance of < or =30 mL/minute at screening, estimated by serum creatinine using the Traub & Johnson equation for calculating pediatric creatinine clearance.

7. a screening BUN or creatinine value that is >1.5 times the upper limit of normal, or liver function tests that are >2 times the upper limit of normal 8. any other screening laboratory test values that the Investigator or Sponsor considers clinically significant that would impact the outcome of the study or the safety of the patient 9. using proton pump inhibitors or antacids 10. pregnant (post-menarchal female patients should be made aware that pregnancy testing will occur during the study, and that if they are sexually active they must take appropriate steps to ensure they do not become pregnant during the study) 11. a positive urine screen for drugs of abuse 12. participated in another clinical trial involving active intervention within 30 days prior to randomization.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | Days 1, 7, 14, 21, and 28

CONTACTS AND LOCATIONS:
Overall Officials: William Aronstein, MD, PhD, Study Director — Procter and Gamble
Locations (22):
- United States (22):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Costa Mesa, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Park Ridge, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Omaha, Nebraska
  - Research Site, Morristown, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Greenville, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Pasadena, Texas
  - Research Site, Seattle, Washington